CLINICAL TRIAL: NCT02367508
Title: Mindfully Optimizing Delivery of End-of-Life Care (MODEL Care): Feasibility of a Synergistic Intervention for Patients, Family Caregivers, and Providers
Brief Title: Mindfully Optimizing Delivery of End-of-Life Care
Acronym: MODEL Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Walther Cancer Institute (Other); Charles Warren Fairbanks Center for Medical Ethics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1312088151
Record Dates: First submitted 2014-12-31; First posted 2015-02-20 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Cancer; Coping Skills
Keywords: advance care planning; coping skills; mindfulness; meditation; cancer; adult; caregivers; oncology providers; advance directives; anxiety; depression; quality of life; pilot project
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MODEL Care (Experimental): Mindfully Optimizing Delivery of End-of-Life Care (MODEL Care) is a mindfulness meditation-based intervention to facilitate timely advance care planning (ACP) and end-of-life conversations with greater ease. Participants are taught a variety of mindfulness practices (e.g., breath awareness, sitting meditation, mindful movement through gentle yoga, and mindful communication) that can be used to enhance end-of-life coping.
  Interventions: Behavioral: MODEL Care

INTERVENTIONS:
Behavioral: MODEL Care — The Mindfully Optimizing Delivery of End-of-Life Care (MODEL Care) intervention is two-pronged and mutually interactive with: (1) a patient and family caregiver group, and (2) an oncology provider group. Patients and family caregivers meet as a group for 6 weekly sessions of 2 hours each, for a total of 12 hours of class time. Oncology providers will have 5 class sessions for a total of 16 hours of class time. One class is held conjointly with patients, family caregivers, and providers to practice newly-learned skills. The course curriculum is generally based on mindfulness practices, group discussion, and didactic teaching with an emphasis on embodying interpersonal mindfulness in dialogue in daily life.

SUMMARY:
The study evaluates the feasibility, acceptability, and preliminary efficacy of a mindfulness meditation-based intervention designed to provide a synergistic solution to the avoidant coping that often inhibits advance care planning discussions that are crucial to quality end-of-life care.

ELIGIBILITY:
Inclusion Criteria:

Oncologists:

* Be a physician specializing in medical oncology
* Care for oncology patients at the affiliated cancer center
* Have a patient panel that will allow for ≥6 eligible patients to be enrolled in the study
* Be willing to attend the 5-session MODEL Care program for providers at the specified location, date, and time

Patients:

* Adults ≥ 18 years of age
* Receiving care from a medical oncologist enrolled in the study
* Diagnosed with an incurable and advanced-stage solid malignancy (late stage III [B or C] or stage IV)
* Have an attending medical oncologist who would not be surprised if the patient died in the next 12 months
* Willing and able to travel to the class location for 6 weekly 2-hour sessions
* Have a family member or friend eligible and interested in participating in the MODEL Care study
* Able and willing to provide informed consent
* Not have completed a Physician Orders for Scope of Treatment (POST) form

Family Caregivers:

* Adults ≥18 years of age
* Chosen by a family member or friend with cancer to join them in participating in the MODEL Care study
* Willing and able to travel to the class location for 6 weekly 2-hour sessions
* Able and willing to consent.

Exclusion Criteria:

Oncologists:

* Planning to leave current practice setting for other employment in the next 3 months.

Patients:

* Eastern Cooperative Oncology Group (ECOG) performance status of >2 or Karnofsky performance status <60 (suggesting patient is capable of only limited self-care, confined to bed or chair more than 50% of waking hours, or requires considerable assistance and frequent medical care) as rated by the attending oncologist
* Currently receiving hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rates at Baseline | Recruitment rates will be estimated at baseline.
  The number of individuals who are eligible will be divided by the number of individuals approached.
Feasibility: Enrollment Rates at Baseline | Enrollment rates will be caluclated at baseline.
  The number of enrolled individuals will be divided by the number of eligible individuals.
Feasibility: Attendance at Post-Intervention (6 weeks) | Attendance will be calculated at the end of the intervention (6 weeks).
  The mean number of sessions attended by each participant type (i.e., patients, family caregivers, providers) will be calculated and compared to the total number of MODEL care sessions provided (i.e., 6 for patients/family caregivers and 5 for providers).
Feasibility: Retention Rates at Post-Intervention (6 weeks) | Retention rates will be calculated at the end of the intervention (6 weeks).
  The proportion of the total number of participants enrolled who completed post-intervention assessments (at 6 weeks) will be calculated by dividing the number of individuals assessed post-intervention (6 weeks) by the number of participants who were enrolled/assessed at baseline.
Acceptability: Intervention Satisfaction at Post-Intervention (6 weeks) | Participants' satisfaction with the intervention will be assessed at the end of the intervention (6 weeks).
  An investigator-created measure of intervention satisfaction will be administered. This measure includes items assessing participants' overall satisfaction, satisfaction with different components of the intervention, likelihood of recommending the course to others, and the intention to continue using MODEL Care skills. The mean score on the satisfaction scale will be calculated for each group (patients, family caregivers, and providers) post-intervention (6 weeks).
Feasibility: Retention Rates at 1-Month Follow-up (10 weeks) | Retention rates will be calculated at 1-month follow-up (10 weeks).
  The proportion of the total number of participants enrolled who completed 1-month follow-up assessments (at 10 weeks) will be calculated by dividing the number of individuals who were assessed at 1-month follow-up (10 weeks) by the number of participants enrolled/assessed at baseline.

SECONDARY OUTCOMES:
Change from Baseline in Avoidant Coping at Post-Intervention (6 weeks) | Avoidant coping will be measured at baseline and post-intervention (6-weeks) for all three groups (patients, family caregivers, and health care providers).
  To measure avoidant coping, the Brief COPE and Mini-Mental Adjustment to Cancer (Mini-MAC) scales will be administered to patients and family caregivers. To assess avoidance among participating health care providers, items adapted from a study assessing effects of end-of-life communication training, and 4 subscales from the Young-Rygh Avoidance Inventory will be used. The effects of MODEL Care on avoidant coping will be determined by calculating the change in avoidant coping scores from baseline to post-intervention (6 weeks) for each group of participants on their respective measures.
Change from Baseline in Avoidant Coping at 1-Month Follow-up (10 weeks) | Avoidant coping will be measured at baseline and at 1-month follow up (10 weeks) for all three groups (patients, family caregivers, and health care providers).
  To measure avoidant coping, the Brief COPE and Mini-Mental Adjustment to Cancer (Mini-MAC) scales will be administered to patients and family caregivers. To assess avoidance among participating health care providers, items adapted from a study assessing effects of end-of-life communication training and 4 subscales from the Young-Rygh Avoidance Inventory will be used. The effects of MODEL Care on avoidant coping will be determined by calculating the change in avoidant coping scores from baseline to 1-month follow-up for each group of participants on their respective measures.
Change from Baseline in Quality of Life at Post-Intervention (6 weeks) | Quality of life will be measured at baseline and post-intervention (6 weeks) for all three groups (patients, family caregivers, and health care providers).
  Patients' quality of life will be measured with the McGill Quality of Life Inventory. Family caregivers' quality of life will be assessed with Caregiver Quality of Life Index-Cancer. Health care providers' quality of life will be assessed using the Professional Quality of Life measure, and Satisfaction with Life scale. The effects of MODEL Care on quality of life will be determined by calculating the change in quality of life scores from baseline to post-intervention (6 weeks) for each group of participants.
Change from Baseline in Quality of Life at 1-Month Follow-up (10 weeks) | Quality of life will be measured at baseline and at 1-month follow-up (10 weeks) for all three groups (patients, family caregivers, and health care providers).
  Patients' quality of life will be measured with the McGill Quality of Life Inventory. Family caregivers' quality of life will be assessed with the Caregiver Quality of Life Index-Cancer. Health care providers' quality of life will be assessed using the Professional Quality of Life measure, and Satisfaction with Life scale. The effects of MODEL Care on quality of life will be determined by calculating the change in quality of life scores from baseline to 1-month follow up for each group of participants.
Change from Baseline in Depression at Post-Intervention (6 weeks) | Depression will be measured at baseline and post-intervention (6 weeks) for all three groups (patients, family caregivers, and health care providers).
  Depression will be assessed for all 3 groups using the 8-item Patient Health Questionnaire depression scale (PHQ-8). The effects of MODEL Care on depression will be determined by calculating the change in PHQ-8 scores from baseline to post-intervention ( 6 weeks) for each group of participants.
Change from Baseline in Depression at 1-Month Follow-up (10 weeks) | Depression will be measured at baseline and at 1-month follow-up (10 weeks) for all three groups (patients, family caregivers, and health care providers).
  Depression will be assessed for all 3 groups using the 8-item Patient Health Questionnaire depression scale (PHQ-8). The effects of MODEL Care on depression will be determined by calculating the change in PHQ-8 scores from baseline to 1-month follow up for each group of participants.
Change from Baseline in Anxiety at Post-Intervention (6 weeks) | Anxiety will be measured at baseline and post-intervention (6 weeks) for all three groups (patients, family caregivers, and health care providers).
  Anxiety will be assessed for all 3 groups using the Generalized Anxiety Disorder scale (GAD-7). The effects of MODEL Care on anxiety will be determined by calculating the change in GAD-7 scores from baseline to post-intervention (6 weeks) for each group of participants.
Change from Baseline in Anxiety at 1-Month Follow-up (10 weeks) | Anxiety will be measured at baseline and at 1-month follow-up (10 weeks) for all three groups (patients, family caregivers, and health care providers).
  Anxiety will be assessed for all 3 groups using the Generalized Anxiety Disorder scale (GAD-7). The effects of MODEL Care on anxiety will be determined by calculating the change in GAD-7 scores from baseline to 1-month follow up for each group of participants.
Change from Baseline in Readiness for Advance Care Planning at Post-Intervention (6 weeks) | Readiness for advance care planning will be measured at baseline and post-intervention (6 weeks) for patients only.
  Patients' readiness to complete 3 advance care planning behaviors (i.e., Physician's Orders for Scope of Treatment form, discussing "goals of care" with their oncologist, and discussing "goals of care" with their family) will be assessed. Responses to these 3 items will indicate the patient's stage of readiness (ranging from pre-contemplation to maintenance) on each behavior. The effects of MODEL Care on advance care planning will be determined by calculating the change in readiness stage category on each behavior from baseline to post-intervention (6 weeks) for patients.
Change from Baseline in Readiness for Advance Care Planning at 1-Month Follow-up (10 weeks) | Readiness for advance care planning will be measured at baseline and at 1-month follow-up (10 weeks) for patients only.
  Patients' readiness to complete 3 advance care planning behaviors (i.e., Physician's Orders for Scope of Treatment form, discussing "goals of care" with their oncologist, and discussing "goals of care" with their family) will be assessed. Responses to these 3 items will indicate the patient's stage of readiness (ranging from pre-contemplation to maintenance) on each behavior. The effects of MODEL Care on advance care planning will be determined by calculating the change in readiness stage category on each behavior from baseline to 1-month follow-up for patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A. Johns, PsyD, Principal Investigator — Indiana University School of Medicine

REFERENCES:
- [Derived] Johns SA, Beck-Coon K, Stutz PV, Talib TL, Chinh K, Cottingham AH, Schmidt K, Shields C, Stout ME, Stump TE, Monahan PO, Torke AM, Helft PR. Mindfulness Training Supports Quality of Life and Advance Care Planning in Adults With Metastatic Cancer and Their Caregivers: Results of a Pilot Study. Am J Hosp Palliat Care. 2020 Feb;37(2):88-99. doi: 10.1177/1049909119862254. Epub 2019 Aug 4. PMID 31378080